CLINICAL TRIAL: NCT04547790
Title: Fiber and Diabetes (FAD) Study: Effect of Psyllium vs. Wheat Dextrin on Glycemic Control and Inflammatory Markers in DM2
Brief Title: A Study to Assess the Effect of Psyllium vs. Wheat Dextrin on Glycemic Control and Inflammatory Markets in Diabetes Mellitus 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen L. Kopecky, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-010612
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Psyllium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psyllium group (Experimental): Subjects will take psyllium once daily for the first three days, then twice daily starting Day 4 until the end of the study.
  Interventions: Dietary Supplement: Psyllium
- Wheat Dextrin group (Experimental): Subjects will take wheat dextrin once daily for the first three days, then twice daily starting Day 4 until the end of the study.
  Interventions: Dietary Supplement: Wheat Dextrin

INTERVENTIONS:
Dietary Supplement: Psyllium — One level scoop (12.5mL) of 5.1g of psyllium fiber twice a day with 8 ounces water
  Other Names: Metamucil
  Arms: Psyllium group
Dietary Supplement: Wheat Dextrin — One level scoop (12.5 mL) of 1.7g wheat dextrin fiber twice a day with 8 ounces water
  Other Names: Benefiber
  Arms: Wheat Dextrin group

SUMMARY:
The purpose of this study is to determine which of Psyllium and Wheat Dextrin is more effective in lowering fasting blood sugar and hemoglobin A1c, and to evaluate the effects they have on laboratory values.

DETAILED DESCRIPTION:
Patients identified as Type 2 diabetics will be identified via Mayo's electronic data system and verified by review of their medical record. Study coordinators will then send invitation letters to patients who meet initial inclusion criteria via mail or through the Mayo Patient Online Services (i.e. patient portal). Recruitment tools used will be flyer, an internet web posting, and a Mayo classified research ad placed in the Mayo classifieds. If patients are interested in participating, they will call or email the study coordinators to set up their baseline visit. Non-responders will be called up to 3 times if no answer. The study coordinator will ask if they received the letter and if they have any questions and if they are interested in participating.

Potential subjects will be screened and consented either digitally or via paper. After consent, the study coordinator will complete the subject's medical history, review concomitant medications, and record vital signs during the baseline visit. Subjects will be randomized and instructed to complete a baseline blood draw, after which they will be given a 3-month supply of study product, a dosing scoop for the product and instructions on taking the assigned study product. They will be assigned to take the study product once daily for the first three days, then twice daily starting Day 4 until the end of the study.

Subjects will be asked to respond to a text message or email message, daily, asking how many doses of study medication they took for that day (0, 1 or 2). The study coordinator will also contact subjects by phone or email to review and reinforce adherence to the protocol if the survey research center identifies subjects who have not responded to text messages within 3 days.

Subjects will meet with study coordinators in person at 4, 8, and 12 weeks or study end to collect vitals, perform a symptom check, review concomitant medications, complete blood draws, and reinforce adherence to protocol.

ELIGIBILITY:
Subject population: This will include adult ECH patients (18 years of age or older) with DM2 who receive their care and diabetic management through Primary Care in Rochester at Mayo Clinic.

Inclusion Criteria:

* Age >18
* May be on oral therapy (including metformin) or insulin
* Most recent HgbA1c level measuring between 6.5 -10 within the last 3 months
* May be on stable (> 4 weeks) statin dose or no statin therapy
* Willing to sign informed consent and stay on current medical regimen
* Does not use regular dietary fiber supplements; has not had any psyllium containing products in the previous 30 days; is willing to refrain from taking any other fiber containing supplement products during the study
* Has not used systemic steroid agents in the last 30 days
* Able to participate fully in all aspects of the study
* Have access and ability to utilize text messaging or email

Exclusion Criteria:

* Unwilling/unable to participate
* Comorbid inflammatory bowel disease, celiac sprue, nephrotic syndrome, severe cholestasis (e.g., primary biliary cirrhosis), or history of bariatric surgery/bowel resection
* Alcohol use in excess of 14 drinks/week
* Allergic reactions to psyllium or wheat dextrin
* Has participated in a clinical drug study or used an investigational new drug during the previous 30 days
* Self-Report of known or suspected pregnancy or immediate plans (within 3 months) of becoming pregnant
* Currently breastfeeding
* Has a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence
* Anticipated or recent major changes in diet or exercise routine
* Anticipated colonoscopy prep during 3 months of study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood sugar | 12 weeks
  The two endpoints of primary interest for this study are HbA1c and fasting glucose. The primary analysis will assess the change in these endpoints between the two treatment groups over the 12 week study period. To estimate the difference between study groups a linear mixed model will be used to account for repeated measures of subjects. The independent variable will be Psyllium group and the baseline outcome result will be included as a covariate.
Change in HbA1c | 12 weeks
  The primary analysis will assess the change in these endpoints between the two treatment groups over the 12 week study period. To estimate the difference between study groups a linear mixed model will be used to account for repeated measures of subjects. The independent variable will be Psyllium group and the baseline outcome result will be included as a covariate.

SECONDARY OUTCOMES:
Change in LDL-C | 12 weeks
  As a secondary analysis, LDL-C, will be collected and analyzed. to determine any difference between the two groups. The blood chemistry labs will be analyzed using a linear mixed model with the given outcome variable included as a covariate.
Change in ceramides | 12 weeks
  As a secondary analysis, ceramides will be collected and analyzed to determine any difference between the two groups. The blood chemistry labs will be analyzed using a linear mixed model with the given outcome variable included as a covariate.
Change in blood pressure | 12 weeks
  Blood pressure will be collected and analyzed. For vital signs measurements a paired t-test will be used to determine any difference between the two groups. The blood chemistry labs will be analyzed using a linear mixed model with the given outcome variable included as a covariate.
Change in weight | 12 weeks
  Weight will be collected and analyzed. For vital signs measurements a paired t-test will be used to determine any difference between the two groups. The blood chemistry labs will be analyzed using a linear mixed model with the given outcome variable included as a covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kopecky, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No